CLINICAL TRIAL: NCT06185868
Title: Clinical Research Plan for Human Myopia Models
Status: Completed | Type: Observational
Sponsor: Robotrak Technologies Co., Ltd. (Industry)
Responsible Party: Sponsor
Other Study IDs: RYMX202201
Record Dates: First submitted 2023-12-05; First posted 2023-12-29 (Actual); Last update posted 2023-12-29 (Actual); Status verified 2023-12

CONDITIONS: Human Myopia Model

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Samples Without DNA
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: No intervention measures — No intervention measures

SUMMARY:
Collect optical biological parameters, refractive index data, and other related parameters of myopia and refractive errors in children and adolescents, and establish an optical model of myopia in children and adolescents.

DETAILED DESCRIPTION:
Experimental research purpose:Collect optical biological parameters, refractive index data, and other related parameters of myopia and refractive errors in children and adolescents, and establish an optical model of myopia in children and adolescents.

Case selection: This study requires the inclusion of children and adolescents aged between 4 and 18 years who have been diagnosed with myopia and refractive errors through medical examination of dilated pupils.

Plan: Collect eye parameters such as refractive power, whole eye aberration, corrected visual acuity, pupil diameter, axial length, anterior and posterior corneal surface curvature, and corneal thickness of all subjects under 9 non dilated stimuli.

ELIGIBILITY:
Selection criteria:

1. Gender unlimited
2. Age 6-16 years old
3. Through medical optometry with dilated pupils, the spherical equivalent refractive index is within the range of -0.5DS~-8.0DS, and the cylindrical lens is ≤ -0.75DC

Exclusion criteria:

1. Patients with corneal diseases such as corneal ulcers, corneal opacities, and corneal leukoplakia
2. Patients with refractive media opacity, such as cataracts and vitreous hemorrhage
3. Glaucoma patients
4. Patients with nystagmus
5. Patients with strabismus and amblyopia
6. Patients with fundus diseases
7. Patients with a column mirror range greater than -0.75DC
8. Patients with binocular anisometropia ≥ 1.0D
9. Corneal contact lenses (such as corneal reshaping lenses, multifocal contact lenses, and RGP) with a history of wearing
10. Long term history of low concentration atropine and other ocular medications
11. Wearing history of functional lenses such as asymptotic multifocal, multi-point myopic defocus, peripheral defocus, etc
12. Patients participating in other eye clinical trials
13. Individuals with mental illness or cognitive impairment who are unable to cooperate

    * Researchers believe that other reasons are not suitable for clinical trial participants, such as poor physical condition on the day of the trial

Ages: 6 Years to 16 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Recruited volunteers
Sampling Method: Non-Probability Sample
Enrollment: 2000 (Actual)
Dates: Start 2022-05-01 (Actual); Primary Completion 2022-10-30 (Actual); Study Completion 2022-10-30 (Actual)

PRIMARY OUTCOMES:
Refraction | 7 months
  Units of measurement:Diopter; measurement tool: subjective refraction;
Whole eye aberration | 7 months
  Units of measurement:micorn; measurement tool: Visual quality analyzer;
Pupil diameter | 7 months
  Units of measurement:millimetre; measurement tool Visual quality analyzer;
Eye axis length | 7 months
  Units of measurement:millimetre; measurement tool: IOLMaster 700(ZEISS)
Corneal anterior and posterior surface curvature | 7 months
  Units of measurement:Diopter; measurement tool: Petacam HR
Corneal thickness | 7 months
  Units of measurement:millimetre; measurement tool: Petacam HR
Anterior Chamber Depth | 7 months
  Units of measurement:millimetre; measurement tool: Petacam HR
Corrected Visual Acuity | 7 months
  Units of measurement:NA; measurement tool: subjective refraction;
Intraocular Pressure | 7 months
  Units of measurement:millimeters of mercury height; measurement tool: Tonometer (NT-510)

CONTACTS AND LOCATIONS:
Locations (1):
- Robotrak Technologies Co., Ltd., Nanjing, China